CLINICAL TRIAL: NCT01445717
Title: Use of a New Rapid Method, BioNanoPore, for Growth and Detection of Group B Streptococcus in Pregnant Patients
Brief Title: Rapid Diagnostic Test for Detection of Group B Streptococcus in Pregnancy
Acronym: GBS
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jonathan P Faro, Assistant Professor, ObGyn, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-10-0317
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Streptococcus Infection; Pregnancy
Keywords: GBS, Streptococcus, .; Group B
MeSH Terms: conditions — Streptococcal Infections; Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens are to be retained for one month, frozen in LIM broth, and will be held for use if reprocessing specimens is required.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the use of a new method of growing and detecting Group B streptococcus in pregnant women. This new method utilizes sandwiched-membrane petri technology and has the advantage of detecting GBS in less than 6 hours, with less cost, and the potential of allowing antibiotic sensitivities to be performed.

DETAILED DESCRIPTION:
Intrapartum infection with group B streptococci (GBS) may lead to untoward neonatal sequelae such as pneumonia, septicemia, and meningitis. Several clinical trials have demonstrated that the use of intrapartum intravenous antibiotic prophylaxis (with penicillin being the agent of choice due to a narrower spectrum of antimicrobial activity) is highly effective to prevent early-onset neonatal GBS infections. It has been estimated that 10% to 30% of all pregnant women are GBS carriers, and it is likely that GBS colonizes virtually every female at some point. Consensus guidelines from the Centers for Disease Control and Prevention (CDC), American College of Obstetricians and Gynecologists (ACOG), and the American Academy of Pediatrics, recommend prenatal screening at 35 to 37 weeks of gestation and chemoprophylaxis at delivery based upon this culture result. The CDC-recommended method for detecting GBS colonization involves collecting a combined vaginal and rectal specimen and culturing the organism in a selective broth medium, followed be subculturing onto blood agar plates.

However, this traditional method of culture takes up to 72 hours for results to be available. With 12.8% of patients experiencing a preterm delivery prior to when a GBS screening occurs, and up to 15% of term pregnancies not having routine GBS screening performed, a significant portion of women present with unknown GBS status at the time of potential delivery. These clinical situations require obstetricians to utilize a risk-based strategy that has been shown to be only half as effective as culture-based screening. Thus, a need exists for a rapid detection method for GBS.

Recent research has focused on polymerase chain reaction (PCR) based methods for detection of GBS. Sensitivity for detection of GBS by the PCR assay has ranged from 87% to 91%. These methods are limited by high cost, and inability to perform antibiotic sensitivities for GBS (in women with a penicillin allergy). New technologies, called bionanopore (BNP) and bionanofilter (BNF) are rapid, microbial detection systems that utilizes sandwiched-membrane petri technology. These have the advantage of detecting GBS in less than 6 hours, with less cost, and the potential of allowing antibiotic sensitivities to be performed.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* 35-37 weeks pregnancy
* Patient receiving prenatal care at UT Houston Hermann Memorial OB/Gyn resident or attending clinic.

Exclusion Criteria:

* Pt elects not to participate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant patients who present to the UT resident or attending clinic between 35-37 weeks for routine follow-up will be asked to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Culture of Group B streptococcus | 48 hours
  Rapid assay results will be compared to routine culture results.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Faro, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UTHSC at Houston, Houston, Texas, United States